CLINICAL TRIAL: NCT06620198
Title: Effects of Robot-Assisted Therapy for Upper Limb Functional Recovery in Patients with Guillain-Barré Syndrome: a Randomized Controlled Trial
Brief Title: Upper Limb Robot-Assisted Therapy in Patients with Guillain-Barré Syndrome
Acronym: RAUL-Project
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110SL24
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-09

CONDITIONS: Guillain Barré Syndrome
Keywords: Polyradiculopathy; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Polyradiculoneuropathy; Exoskeleton device; Robotic Rehabilitation
MeSH Terms: conditions — Guillain-Barre Syndrome; Polyradiculopathy; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Polyradiculoneuropathy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors, Patients and their caregivers will be blinded for the entire duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active-assisted therapy with an upper limb robotic exoskeleton (Experimental): Patients will receive upper limb neurorehabilitation training using a robotic exoskeleton administered by the therapist. The assistance provided by the device is adjusted based on the maximum force (as a percentage of the upper limb's weight) the robot needs to exert to assist the patient's movements. The computer-robot interface is designed to offer various exergames that require specific upper limb movements.
  All movements performed by the patient using the exoskeleton will provide immediate audiovisual feedback on the computer screen. The training will consist of 20 sessions, with five 45-minute sessions per week.
  Interventions: Device: Armeo® Power 2 Exoskeleton - Active Rehabilitation with Feedback and Exercise Gaming
- Passive mobilization with an upper limb robotic exoskeleton (Active Comparator): Patients will undergo a neurorehabilitation intervention with a SHAM treatment under the guidance of the experimental therapist.
  Interventions: Device: Armeo® Power 2 Exoskeleton - Passive Mobilization without Feedback

INTERVENTIONS:
Device: Armeo® Power 2 Exoskeleton - Active Rehabilitation with Feedback and Exercise Gaming — Patients will undergo 20 session of 45 minutes each with an exoskeleton for upper limb rehabilitation. The assistance provided by the device is adjusted based on the maximum force (as a percentage of the upper limb's weight) the robot needs to exert to assist the patient's movements. Each session will include exercises designed to improve the range of motion (ROM) of the shoulder, elbow, wrist, and enhance hand coordination. The training parameters, such as difficulty level, duration, and visual stimuli, will be adjusted based on the patient's residual abilities. The selected exercises may involve movements of a single joint along one axis, combined movements of a single joint around 2 or 3 axes, selective exercises for the opening and closing hand, or multi-joint exercises. All exercises will be realized with audiovisual feedback.
  Arms: Active-assisted therapy with an upper limb robotic exoskeleton
Device: Armeo® Power 2 Exoskeleton - Passive Mobilization without Feedback — Patients will undergo 20 session of 45 minute of a neurorehabilitation intervention with a SHAM treatment under the guidance of the experimental therapist. This will involve passive mobilization using the exoskeleton for the upper limb, without any audiovisual feedback. They will not realize any active movement during the training.
  Arms: Passive mobilization with an upper limb robotic exoskeleton

SUMMARY:
Guillain-Barré Syndrome is an immune-mediated polyradiculoneuropathy, with around 100,000 new cases reported worldwide annually.

The aim of this double-blind randomized controlled trial with a SHAM control group is to evaluate the effects of robot-assisted therapy, integrated with conventional therapy, on upper limb motor recovery in patients with GBS.

DETAILED DESCRIPTION:
Guillain-Barré Syndrome is a leading cause of acute flaccid paralysis, presenting with limb weakness and hyporeflexia or areflexia. Guillain-Barré Syndrome is an immune-mediated polyradiculoneuropathy, with around 100,000 new cases reported worldwide annually. This study aims to assess the effectiveness of a robot-assisted rehabilitation treatment for upper limb motor recovery in patients with Guillain-Barré Syndrome. A double-blind randomized trial will be conducted, where the experimental group will undergo actual robotic rehabilitation sessions, while the control group will perform sessions in which the robot will carry out simple mobilization, comparable to traditional interventions. This approach will help maintain participant blinding. Patients will be evaluated before and after treatment, and with two follow-up assessments 60 and 90 days after therapy initiation. Evaluations will include muscle recruitment and autonomy in daily living activities.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Guillan-Barré Syndrome;
2. UL motor impairment (0-4 in the Medical Research Council scale);
3. sub-acute phase (until 180 days);
4. Patients able to maintain the sitting position.

Exclusion Criteria:

1. Concomitant neurological, orthopedic, metabolic, and oncological diseases;
2. Cognitive impairment assessed with the Mini Mental State Examination (score under 24 points);
3. Visual deficit;
4. Hearing disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment scale for Upper Extremity (FMAUE) | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  THE FMAUE will be used to assess the change in the motor and sensory functions of the upper limb. The FMAUE included five domains: motor functioning, sensitivity, coordination, range of motion and pain. The score ranging from 0 to 66 points, a higher score corresponds to a better function of the upper limb.

SECONDARY OUTCOMES:
The 36-Item Short-Form Health Survey (SF-36) | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  The SF-36 will be used to assess the change in health-related quality of life. The SF-36 is organized into 8 different domains that are divided into physical components (Physical functioning, limitations due to physical problems, bodily pain and general perceptions of health status) and mental components (Social functioning, general mental health, limitations due to emotional problems and vitality). Each of the 8 domain scores, added together, is linearly transformed on a scale from 0 to 100, where 0 equals negative health and 100 equals positive health.
modified Barthel Index (mBI) | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  The mBI will be used to assess the change in the autonomy of patients during their activities of daily living. This scale has a score ranging from 0 to 100 points, a higher score corresponds to a better performance in the activities of daily living.
ABILHAND | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  The ABILHAND will be used to assess manual dexterity. The ABILHAND is a questionnaire-based assessment tool that measures the difficulty a patient perceives in using their hands to perform manual operations and activities in daily living. It assesses upper limb functionality. It has nonlinear logit values ranging from 1.72 to -2.18.
The Medical Research Council scale (MRC) | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  The MRC will be used to assess muscle strength. The score ranges from 0 to 5 where 0 equals no muscle recruitment and 5 normal muscle force.
The nine hole peg test (NHPG). | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  The NHPG will be used to assess fine manual dexterity. The NHPT consists of a square board with 9 pegs. At one end of the board are holes to insert the pegs, and at the other end is a shallow round plate to store the extracted pegs. The NHPT is administered by asking the patient to take the pegs from a container, one by one, and insert them into the holes on the board, as quickly as possible.
Grip strength | Baseline (t0); 30 days (t1); 60 days (t2); 90 days (t3).
  Grip strength will be assessed using a manual digital dynamometer. The maximum strength of the whole hand will be recorded for three times without feedback (with the patient sitting with his back to the monitor).

OTHER OUTCOMES:
Mini-Mental State Examination (MMSE) | T0 (Baseline)
  MMSE is a widely used psychometric tool in clinical settings to assess cognitive function. It is employed to detect cognitive impairments, monitor the progression of neurodegenerative diseases such as Alzheimer disease, and evaluate the severity of cognitive decline.
  The test consists of a series of questions and tasks that assess various cognitive domains, including orientation in time and space, memory, attention, language, and the ability to follow simple commands.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Martino Cinnera, PhD, Study Chair — IRCCS Santa Lucia Foundation; Diego Piatti, BSc, Study Chair — IRCCS Santa Lucia Foundation; Laura Casagrande Conti, MSc, Study Director — IRCCS Santa Lucia Foundation; Martina D Arienzo, BSc, Study Director — IRCCS Santa Lucia Foundation
Locations (1):
- IRCCS Santa Lucia Foundation, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2024/10/01
Access Criteria: on resonable request to the study' PI